CLINICAL TRIAL: NCT06092853
Title: Inflammatory Stress and Periodontal Tissue Destruction in Patients With Metabolic Syndrome and Periodontitis
Brief Title: Inflammatory Stress and Periodontal Tissue Destruction
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Collaborators: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Hatice Yemenoğlu, assistant professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: Recep Tayyip ErdoganUniversity; RecepTayyipErdoganUniversity (Other: Recepteutrh)
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Oxidative Stress; Inflammation
Keywords: Metabolic syndrome; periodontitis; interleukin-20
MeSH Terms: conditions — Inflammation; Metabolic Syndrome; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — plasma and gingival crevicular fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- systemically and periodontally healthy (CG): Gingival crevicular fluid (GCF) and serum samples were collected from all participants for biochemical analyses.
  Interventions: Other: Gingival crevicular fluid (GCF) and serum samples
- systemically healthy and periodontitis (PG): Gingival crevicular fluid (GCF) and serum samples were collected from all participants for biochemical analyses
  Interventions: Other: Gingival crevicular fluid (GCF) and serum samples
- Metabolic syndrome and periodontally healthy (MG): Gingival crevicular fluid (GCF) and serum samples were collected from all participants for biochemical analyses
  Interventions: Other: Gingival crevicular fluid (GCF) and serum samples
- Metabolic syndrome and periodontitis (MPG): Gingival crevicular fluid (GCF) and serum samples were collected from all participants for biochemical analyses
  Interventions: Other: Gingival crevicular fluid (GCF) and serum samples

INTERVENTIONS:
Other: Gingival crevicular fluid (GCF) and serum samples — Gingival crevicular fluid (GCF) and serum samples were collected from all participants for biochemical analyses

SUMMARY:
Metabolic syndrome and periodontitis are diseases that lower the quality of life and their incidence rates are increasing. Since both of these diseases are associated with systemic inflammation and insulin resistance, they may be comorbid. The aim of this study was to evaluate the effect of interleukin-20 (IL-20) on periodontal destruction in individuals with metabolic syndrome while considering the relationship between metabolic syndrome and periodontitis.

This study included a total of 80 individuals who were systemically and periodontally healthy (CG, n=20), were systemically healthy and had periodontitis (PG, n=20), had metabolic syndrome and were periodontally healthy (MG, n=20), or had both metabolic syndrome and periodontitis (MPG, n=20). Gingival crevicular fluid (GCF) and serum samples were collected from all participants for biochemical analyses.

ELIGIBILITY:
Study groups were created based on the guidelines of the 2017 Classification of Periodontal Diseases and the 2005 Metabolic Syndrome Diagnostic Criteria of the Endocrinology and Metabolic Society of Turkey

Inclusion Criteria:

* all participants were required to have at least 20 teeth and be between the ages of 20 and 65 years

Exclusion Criteria:

* Smokers, patients who had used antibiotics or anti-inflammatory and antioxidant drugs in the last 6 months, patients who were pregnant or lactating, those who had cancer or autoimmune diseases, and those who had undergone any periodontal treatment in the last 6 months

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size of the study was calculated using the G*Power program with an effect size of 0.4, 80% power, and a margin of error of 0.05.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
concentration of gingival crevicular fluid (GCF) parameters | 1 year
  interleukin-20, RANKL, OPG values evaluated in GCF.
concentration of serum parameters | 1 year
  interleukin-20, RANKL, OPG, MMP-8, TOS, TAS values evaluated in serum

SECONDARY OUTCOMES:
value of periodontal clinical parameters | 1 year
  plaque index, gingival index, bleeding on probing, Clinical attachment loss, probing pocket depth
value of patients' clinical metabolic syndrome parameters | 1 year
  Body mass index (BMI), abdominal circumference, and HbA1c

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdogan University, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Senkal R, Yemenoglu H, Kose O, Karakas SM, Yilmaz A, Akyildiz K, Beder M, Bostan SA. The role of interleukin-20 on inflammatory stress and periodontal tissue destruction in patients with metabolic syndrome and periodontitis. BMC Oral Health. 2024 Nov 22;24(1):1423. doi: 10.1186/s12903-024-05224-3. PMID 39578819